CLINICAL TRIAL: NCT05374863
Title: Evaluation and Intervention of Intradialytic Physical Therapy in Patients With Chronic Kidney Disease: a Randomized Clinical Trial Protocol
Brief Title: Intradialytic Physiotherapy in Patients With Chronic Kidney Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Marcela Cangussu Barbalho (Other)
Collaborators: Hospital Universitário Cassiano Antônio Moraes (Unknown)
Responsible Party: Sponsor-Investigator, Marcela Cangussu Barbalho, Principal Investigator, Federal University of Espirito Santo
Organization: Federal University of Espirito Santo (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 27067819.1.0000.5071
Record Dates: First submitted 2022-04-12; First posted 2022-05-16 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Chronic Renal Diseases
Keywords: Chronic kidney disease; Hemodialisis; Exercise; Neuromuscular electrical stimulation
MeSH Terms: conditions — Renal Insufficiency, Chronic; Motor Activity

STUDY DESIGN:
Intervention Model Description: This is a controlled, randomized, double-blind clinical trial with an intention-to-treat analysis.
Who Masked: Participant, Outcomes Assessor
Masking Description: This is a double-blind study, where evaluators and participants will not be aware of the details of the research. All outcomes will be measured by blinded raters as they will not be involved in the randomization process and will not receive details about interventions. All participants will be blinded as to whether or not the NMES will be performed, as both the intervention group and the control group will have the electrodes positioned and will remain there for the same time.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Neuromuscular electrical stimulation (NMES) active in the upper limbs for 20 minutes and aerobic exercises on the cycle ergometer for 30 minutes.
  Interventions: Device: Neuromuscular electrical stimulation (NMES) - Active; Device: Aerobic exercise with cycle ergometer
- Control Group (Placebo Comparator): NMES-Sham in upper limbs for 20 minutes and aerobic exercises on a cycle ergometer for 30 minutes.
  Interventions: Device: Neuromuscular Electrical Stimulation (NMES) - Sham; Device: Aerobic exercise with cycle ergometer

INTERVENTIONS:
Device: Neuromuscular electrical stimulation (NMES) - Active — The NMES will be held for 20 minutes. Biceps musculature and bilateral wrist and finger flexors stimulated. For patients undergoing hemodialysis for fistula in the upper limb, NMES will be performed only in the limb without a fistula. points of points 4 electrodes in each, being 2 points of longitudinal position in the muscular belly of the biceps, and other 2 in the ventral region of the forearm. the parameters: frequency of 80 Hz, pulse frequency of 350 ms, time of 5 seconds and 10 seconds. The possibility will be greater for each patient who will have the contraction. Patients will be instructed to perform an isometric contraction of wrist and finger flexors during electrical stimulation.
  Arms: Experimental Group
Device: Neuromuscular Electrical Stimulation (NMES) - Sham — It will be performed in the same way as in the experimental group, however, the intensity of the actuality will only reach the sensitive threshold.
  Arms: Control Group
Device: Aerobic exercise with cycle ergometer — The exercise will be performed from the adaptation and positioning of a cycle ergometer (Mini Bike E5 Acte Sports®) in front of the hemodialysis chair. Each session will consist of three phases: duration (5 minutes), conditioning (20 minutes) and cool-down (5 minutes). During the development and cool-down phases, patients will be instructed to maintain a lower exercise intensity, with a level between 1 and 3 on the modified BORG scale. In the conditioning phase, patients will be instructed to slightly increase the intensity of the exercise, levels between 4 and 7 on the modified BORG scale. During exercise, patients will be asked every 5 minutes about the level of effort, and the load on the cycle ergometer will be possible to reach an intensity between 4 and 7 on the modified Borg Scale.

SUMMARY:
The objective is to evaluate in adult patients with chronic kidney disease the effect of neuromuscular electrical stimulation (NMES) in the upper limbs associated with a cycle ergometer in the lower limbs, during hemodialysis, on functional capacity and peripheral muscle strength.

The hypothesis is that in people with chronic kidney disease on hemodialysis, the addition of neuromuscular electrical stimulation in the upper limbs associated with aerobic training of the lower limbs is superior to aerobic exercise alone in improving functional capacity, peripheral muscle strength, quality of life, safety intervention and patient adherence.

DETAILED DESCRIPTION:
Objective: To evaluate, in adult patients with chronic kidney disease, the effect of neuromuscular electrical stimulation (NMES) in the upper limbs associated with a cycle ergometer in the lower limbs, during hemodialysis, on functional capacity and peripheral muscle strength.

Methods. This is a controlled, randomized, double-blind, intention-to-treat clinical trial carried out at the Cassiano Antônio Moraes University Hospital (HUCAM). Thirty individuals who will be randomly allocated to an intervention group (ie active NMES on upper limbs for 20 minutes and aerobic exercise on a cycle ergometer for 30 minutes) or a control group (ie NMES-Sham on upper limbs for 20 minutes and aerobic exercise on a cycle ergometer for 30 minutes). The treatment will be carried out for 8 weeks, with 3 weekly sessions totaling 24 sessions. Outcome measures will be collected by trained researchers before treatment (week 0) and at the end of treatment (week 9), always in the second hemodialysis session of the week. Functional capacity, peripheral muscle strength, activity level of daily living, quality of life, intervention safety, patient compliance, hemodialysis filtration rate (KT/V) and renal function (potassium, phosphate and magnesium clearance) will be evaluated.

Impact. This study could potentially provide important information and assist in clinical decision making regarding the combined use of NMES with a cycle ergometer to optimize the clinical benefits of therapeutic exercise in patients with chronic kidney disease.

ELIGIBILITY:
Inclusion Criteria:

* Have chronic kidney disease;
* Undergo hemodialysis at HUCAM for at least 3 months;
* Present a hemoglobin level > 9 g/dL;
* Present clinical stability for at least 3 months;
* Do not participate in another physical exercise program;
* Present the ability to perform the assessment tests;
* Age equal to or greater than 18 years, and can be of both sexes;
* Accept to participate in the research by signing the informed consent form.

Exclusion Criteria:

* Presents symptoms and/or health conditions (cardiovascular, respiratory, neurological, cognitive) that prevent the performance of evaluation tests and participation in the exercise program.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Improved Functional Capacity | Baseline, pre-intervention/immediately after intervention.
  It will be evaluated by the one-minute sit-and-stand test. Patients will be instructed to sit and stand up in a chair as quickly as possible for 1 minute, starting from the sitting position, with their feet on the floor, arms crossed on the chest and back supported on the chair, in addition, they will not receive any type of incentive verbal during the test. The number of repetitions will be recorded, and if the participant is standing at the end of 1 minute, 0.5 repetition will be considered.
Improved Peripheral muscle strength | Baseline, pre-intervention/immediately after intervention.
  It will be evaluated through the handgrip strength being measured using a manual digital dynamometer (Instruthern®, São Paulo, Brazil). The test will be performed three times on each upper limb (right and left), with 1-minute intervals between each execution, the measure with the highest value being considered.

SECONDARY OUTCOMES:
Improved Cardiorespiratory capacity | Baseline, pre-intervention/immediately after intervention.
  It will be evaluated through the self-administered questionnaire called Duke Activity Status Index (DASI), which is composed of 12 items covering personal care, household activities, sexual activity and recreational activities. Item scores are graded based on metabolic cost measured in metabolic equivalents (METs). Each item with the answer "YES" receives a score ranging from 1.75 to 8.00 points. "NO" answers are scored as 0. The total score ranges from 0 to 58.2 points, with higher scores meaning greater cardiorespiratory capacity. From the result of the sum of the scores of the 12 items, it is possible to estimate the oxygen consumption at the peak of the exercise (VO2peak), since a strong correlation between the DASI and the VO2peak obtained from the cardiopulmonary test (gold standard) has already been demonstrated.
Improved Capacity of life. | Baseline, pre-intervention/immediately after intervention.
  It will be evaluated using the Kidney Disease and Quality of Life Short-Form (KDQOL-SFTM) questionnaire, which is a specific instrument that assesses the quality of life in patients with end-stage renal disease, applicable to patients undergoing some type of dialysis program. . It is a self-administered instrument with 80 items, divided into 19 scales. It is a complete questionnaire, as it includes generic and specific aspects related to kidney disease.

CONTACTS AND LOCATIONS:
Overall Officials: Marcela c Barbalho, PhD, Principal Investigator — Federal University of Espírito Santo
Locations (1):
- Federal University of Espírito Santo, Vitória, Espírito Santo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rosa MR, de Souza VS, Paro FM, Gomes DCAP, Toledo MLSA, Pedreira AB, Duarte H, Wittmer VL, Moulim MCB. Safety and Feasibility of Intradialytic Exercise Including Upper Limb Neuromuscular Electrical Stimulation in Adults With Chronic Kidney Disease: A Randomized Controlled Pilot Clinical Trial. Artif Organs. 2025 Aug 13. doi: 10.1111/aor.70006. Online ahead of print. PMID 40799154
- See also: A brief self-administered questionnaire to determine functional capacity (the Duke Activity Status Index). — https://doi.org/10.1016/0002-9149(89)90496-7
- See also: Translation and cross-cultural adaptation of the Duke Activity Status Index to Brazilian Portuguese. — https://doi.org/10.1590/S0103-51502013000300017
- See also: Tradução e adaptação cultural do instrumento de avaliação de qualidade de vida para pacientes renais crônicos (KDCOL-SFTM). — https://doi.org/10.1590/S0104-42302003000400027
- See also: Development of the kidney disease quality of life (KDQOL) instrument. — https://doi.org/10.1007/BF00451725
- See also: Brazilian Dialysis Census: analysis of data from the 2009-2018 decade. — https://doi.org/10.1590/2175-8239-JBN-2019-0234
- See also: Efeito da estimulação elétrica neuromuscular na força muscular, capacidade funcional e composição corporal em pacientes em hemodiálise. — https://doi.org/10.1016/j.nefro.2016.05.010
- See also: A carga global da doença renal crônica. — https://doi.org/10.1016/S0140-6736(19)32977-0
- See also: Diretrizes de Prática Clínica para o Manejo da Pressão Arterial na Doença Renal Crônica — https://doi.org/10.1016/j.kint.2020.11.003